CLINICAL TRIAL: NCT04640428
Title: COVID-19 Stroke Apical Lung Examination Study - A Multi-centre Prospective Study
Brief Title: COVID-19 Stroke Apical Lung Examination Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVID SALES 2
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Stroke, Acute; Stroke, Ischemic; Stroke Hemorrhagic
Keywords: COVID; stroke; CT; CTA
MeSH Terms: conditions — COVID-19; Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multi-centre prospective study evaluating computed tomography angiography studies performed for stroke patients as a diagnostic and prognostic imaging biomarker.

DETAILED DESCRIPTION:
Diagnosis of coronavirus disease 2019 (COVID-19) relies on clinical features and reverse-transcriptase polymerase chain reaction (RT-PCR) testing. The latter is constrained by limited sensitivity and a timescale of hours to yield results, with no point-of-care test widely available. A dedicated computed tomography study of the chest is likely to be more sensitive than RT-PCR for COVID-19. Carotid computed tomography angiography (CTA) is a routine acute stroke investigation and includes the lung apices. We aim to assess the lung apices on CTA for ground glass opacification and compare this with COVID-19 RT-PCR test results and clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

All adult patients presenting with clinical features of acute ischaemic stroke undergoing investigation with computed tomography angiography at presentation.

Exclusion Criteria:

Poor image quality. No radiologist report available. Computed tomography angiography performed in a non-acute setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to participating centres with clinical features of acute ischaemic stroke undergoing investigation with computed tomography angiography at presentation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the computed tomography angiography biomarker relative to the COVID-19 RT-PCR test | 1 month
  Defined by sensitivity, specificity, positive and negative predictive values

SECONDARY OUTCOMES:
Prognostic value of the computed tomography biomarker | 1 month
  Defined by its relationship with 30 day mortality and modified rankin scale following treatment

CONTACTS AND LOCATIONS:
Locations (12):
- United Kingdom (12):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - North Bristol NHS Trust, Bristol
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Frimley Health NHS Foundation Trust, Camberley
  - Cardiff and Vale University Health Board, Cardiff
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Foundation Trust, London
  - King's College Hospital NHS FT (KCH), London
  - King's College Hospital NHS FT (PRUH), London
  - University College London NHS Foundation Trust, London